CLINICAL TRIAL: NCT07000695
Title: Managed Access Programs for TQJ230, Pelacarsen
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTQJ230A12013M
Record Dates: First submitted 2025-05-12; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Atherosclerotic Cardiovascular Disease, ASCVD
Keywords: MAP; Manage Access Program; TQJ230; Pelacarsen; Atherosclerotic Cardiovascular Disease; ASCVD
MeSH Terms: conditions — Atherosclerosis | interventions — pelacarsen

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Pelacarsen — Patients receive Pelacarsen
  Other Names: TQJ230

SUMMARY:
The purpose of this registration is to list Managed Access Programs (MAPs) related to TQJ230, pelacarsen

DETAILED DESCRIPTION:
CTQJ230A12013M - Available - Managed Access Program (MAP) Cohort Treatment Plan (CTQJ230A12013M) to provide access to pelacarsen (TQJ230) for (Atherosclerotic Cardiovascular Disease, ASCVD)

ELIGIBILITY:
Inclusion Criteria:

1. An independent request was received from a licensed physician.
2. The patient has a serious or life-threatening disease or condition and there is no comparable or satisfactory alternative therapy available for diagnosis, monitoring, or treatment.
3. The patient is not eligible or able to enrol in a clinical trial or continue participation in such trial.
4. There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated.
5. The patient must meet any other medical criteria established by the medical experts responsible for the product or by the health authority in the country of request (as applicable).
6. Provision of the product will not interfere with the initiation, conduct, or completion of a Novartis clinical trial or overall development program.
7. Managed Access provision is allowed per local laws/regulations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult